CLINICAL TRIAL: NCT07215468
Title: A Phase 2b Study of the Safety, Pharmacokinetics, and Efficacy of the Combination of TMB-365 and TMB-380 as Maintenance Therapy in HIV-1 Infected Individuals Suppressed With Combination Antiretroviral Therapy
Brief Title: HIV-1 Virologic Suppression With TMB-365 and TMB-380 Antibodies Study
Acronym: VISTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMB-b21
Record Dates: First submitted 2025-10-09; First posted 2025-10-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: HIV -1 Infection
Keywords: HIV-1 maintenance treatment; HIV switch therapy; Broadly neutralizing antibody (bNAb); HIV post-attachment inhibitor; monoclonal antibody (mAb)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination of TMB-365 and TMB-380 antibodies via IV infusions (Experimental): Participants will receive an IV infusion of the combination of TMB-365 and TMB-380 each every 8 weeks.
  Interventions: Drug: TMB-365; Drug: TMB-380
- Baseline oral cART (Active Comparator): Participants will continue suppressive daily oral cART
  Interventions: Drug: Baseline ART

INTERVENTIONS:
Drug: TMB-365 — A monoclonal antibody acts as a HIV post-attachment inhibitor to be given intravenously
  Arms: Combination of TMB-365 and TMB-380 antibodies via IV infusions
Drug: TMB-380 — A broadly neutralizing antibody (bNAb) against HIV to be given intravenously
  Other Names: VRC07-523LS
  Arms: Combination of TMB-365 and TMB-380 antibodies via IV infusions
Drug: Baseline ART — Baseline ART to be taken daily and orally
  Arms: Baseline oral cART

SUMMARY:
TMB-365 is a monoclonal antibody that binds to the CD4 receptor. TMB-380, aka VRC07-523LS is a monoclonal antibody that binds to HIV. Both interfere with HIV entry. This study is designed to test the combination of the antibodies as maintenance therapy in HIV infected suppressed individuals discontinuing oral cART for 48 weeks.

Researchers will compare TMB-365/TMB-380 given IV every 8 weeks to continuation of daily oral cART to see if TMB-365/TMB-380 can also maintain viral suppression.

Participants will:

1. Receive TMB-365/TMB-380 infusion or take oral cART as scheduled for 48 weeks
2. Visit the clinic as schedule for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of Screening.
2. Asymptomatic HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by Geenius™ or a second antibody test by a method other than the initial rapid HIV and/or E/CIA test, or by HIV-1 antigen, plasma HIV-1 RNA viral load at or prior to screening.
3. On continuous suppressive cART for at least 6 months prior to Screening with one documented HIV-1 RNA level <50 copies/mL within 6 months of Screening. Continuous cART is defined as no interruptions greater than 3 consecutive days. cART is defined as a DHHS recommended regimen. Study participants should be on a stable oral regimen for at least 3 months prior to Screening.
4. Screening plasma HIV-1 RNA < 50 copies/mL
5. CD4+ T cell count >350 cells/mm3
6. Laboratory values obtained within 35 days prior to the first dose:

   * Hemoglobin ≥ 10.0 g/dL
   * Platelet count ≥ 100,000/mm3
   * Absolute neutrophil count ≥ 1,000/mm3
   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x upper limit of normal (ULN)
   * Creatinine clearance (CrCl) of ≥ 50 mL/min
7. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
8. In the opinion of the principal investigator or designee, has understood the information provided; written informed consent needs to be given before any study-related procedures are performed.
9. Persons of childbearing potential sexually active with a partner who can impregnate them, must agree to use one effective method of contraception from the time of signing the consent to completion of the study, and agree to pregnancy testing as per the Schedule of Events and Procedures. Persons of childbearing potential are participants born female who are not surgically sterile (no history of bilateral tubal ligation, hysterectomy, or bilateral salpingo-oophorectomy), are not postmenopausal (at least one year without menses), and are not otherwise sterile by medical evaluation.

Exclusion Criteria:

1. Receipt of any monoclonal antibody for the treatment or prevention of HIV infection.
2. Receiving cabotegravir and rilpivirine intramuscularly as maintenance therapy for HIV-1 infection.
3. Pregnant, planning a pregnancy during the trial period, or lactating.
4. Known allergy/sensitivity or any hypersensitivity to components of the study drug or its formulation, or known allergy to a MAb.
5. History of severe allergic reactions to medications, vaccinations, or monoclonal antibody therapy for other conditions such as COVID.
6. Major psychiatric illness including any history of schizophrenia or severe psychosis, uncontrolled bipolar disorder requiring acute therapy, or suicide attempt in the previous three years.
7. Serious illness requiring systemic treatment and/or hospitalization within 21 days prior to Baseline.
8. Receipt of immunomodulatory agents (e.g., interleukins, interferons, cyclosporine, high dose systemic corticosteroids), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 180 days prior to Baseline.
9. Any chronic or acute medical condition, including chronic Hepatitis B infection, chronic Hepatitis C infection with viremia, drug use and alcohol abuse, which in the opinion of the investigator would interfere with evaluation of the study drug.
10. Lack of adequate venous access.
11. Individuals who have experienced virologic failure during treatment with two or more cART treatment regimens and those being treated with regimens containing either ibalizumab, enfuvirtide, maraviroc, or fostemsavir. Note that a change in treatment regimen for intolerance does not meet criteria for treatment failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Antiviral activity of TMB-365 and TMB-380 as maintenance therapy compared to daily oral cART | Week 48
  % of subjects with plasma HIV-1 RNA greater than or equal to 50 c/mL at week 48 by snapshot analysis as defined by US FDA

SECONDARY OUTCOMES:
Number of participants who experience protocol-defined virologic failure | 48 weeks
  Virologic failure is defined as two consecutive plasma HIV-1 RNA levels ≥200 copies/mL obtained at least 2 weeks apart.
Pharmacokinetic profile of TMB-365 | Week 48
  Mean trough concentrations for TMB-365 in Experimental Arm
Pharmacokinetic profile of TMB-380 | Week 48
  Mean trough concentrations for TMB-380 in Experimental Arm
Safety of maintenance treatment regimen | 48 weeks
  Number of participants experience grade 3, grade 4, or serious adverse reactions related study treatment.
Immune effects of maintenance therapy | 48 weeks
  Changes in CD4+ cell counts (cells/mm3) from baseline to Week 48

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Long Beach Education and Research Consultants, Long Beach, California
  - Quest Clinical Research, San Francisco, California
  - CAN Community Health Fort Lauderdale, Fort Lauderdale, Florida
  - Midway Immunology and Research Center (MIRC), Ft. Pierce, Florida
  - CAN Community Health Miami Gardens, Miami Gardens, Florida
  - Midland Medical, Oakland Park, Florida
  - Orlando Immunology Center, Orlando, Florida
  - CAN Community Health Sarasota, Sarasota, Florida
  - Mercer University, Department of Internal Medicine, Clinical Research, Macon, Georgia
  - CAN Community Health Las Vegas, Las Vegas, Nevada
  - The Crofoot Research Center, Inc., Houston, Texas

IPD SHARING:
Plan to Share IPD: No